CLINICAL TRIAL: NCT01660867
Title: Nebulized 3% Hypertonic Saline in the Treatment of Acute Bronchiolitis in the Emergency Department
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: there was no eligible patients
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Hee Lee, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bronchiolitis_1
Record Dates: First submitted 2012-08-03; First posted 2012-08-09 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Acute Bronchiolitis
Keywords: hospital admission within 7 days of 3% NaCl nebulizer vs dexamethasone
MeSH Terms: interventions — Sodium Chloride; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 0.9% saline + oral placebo (Placebo Comparator): nebulized epinephrine + 0.9% saline + placebo => epinephrine + 0.9% saline
  Interventions: Drug: 0.9% saline + oral dexamethasone
- 3% saline + oral placebo (Experimental): nebulized epinephrine + 3% saline + placebo => nebulized epinephrine + 3% saline
  Interventions: Drug: 3% saline + oral placebo
- 0.9% saline + oral dexamethasone (Active Comparator): nebulized epinephrine + 0.9% saline + dexamethasone => nebulized epinephrine + 0.9% saline
  Interventions: Drug: 0.9% saline + oral dexamethasone

INTERVENTIONS:
Drug: 3% saline + oral placebo — nebulized epinephrine + 3% saline + placebo => nebulized epinephrine + 3% saline
  Arms: 3% saline + oral placebo
Drug: 0.9% saline + oral dexamethasone — nebulized epinephrine + 0.9% saline + dexamethasone => nebulized epinephrine + 0.9% saline
  Arms: 0.9% saline + oral dexamethasone; 0.9% saline + oral placebo

SUMMARY:
This is a prospective, randomized, controlled, double-blinded, clinical trial

Subject : 3mo ~ 24mo. aged infants with bronchiolitis

The effect of 3 % NaCl nebulizer or dexamethasone on admission rate of these infants in ED.

DETAILED DESCRIPTION:
Randomly assigned to one of three groups

* Group I : nebulized epinephrine + 0.9% saline + placebo
* Group II : nebulized epinephrine + 3% saline + placebo
* Group III : nebulized epinephrine + 0.9% saline + dexamethasone

Group I received two treatments of nebulized epinephrine mixed 0.9% saline and a total of six oral doses of placebo, group II received nebulized epinephrine mixed 3% saline and oral placebo, and group III received nebulized epinephrine mixed 0.9% saline and oral dexamethasone.

The primary outcome is hospital admission within 7 days after the day of enrollment

ELIGIBILITY:
Inclusion Criteria:

* 3mo ~ 24mo aged patients with bronchiolitis visit to emergency departments
* RDAI score 4-15

Exclusion Criteria:

* < 3mo, > 24mo
* infants who had received oral or inhaled corticosteroids during the preceding 2 weeks
* infants with a previous episode of wheezing or a diagnosis of asthma
* any chronic cardiopulmonary disease
* immunodeficiency
* infants needed intubation
* infants with a previous history of apnea or intubation
* infants with side effect of dexamethasone
* infants born at less than 37 weeks of gestation who had a corrected age of less than 6 weeks at presentation

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
hospital admission within 7 days after the day of enrollment | within 7 days
  hospital admission within 7 days after the day of enrollment(the initial visit to the emergency department)

SECONDARY OUTCOMES:
RDAI score | baseline, between nebulizer, 60min, 120min, 180min, 240min
  RDAI score
respiratory rate | baseline, between nebulizer, 60min, 120min, 180min, 240min
  respiratory rate
Heart rate | baseline, between nebulizer, 60min, 120min, 180min, 240min
  Heart rate
Oxygen saturation | baseline, between nebulizer, 60min, 120min, 180min, 240min
  Oxygen saturation
unplanned revisit and admission rate after revisit | in 7days
  unplanned revisit admission rate after revisit

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea